CLINICAL TRIAL: NCT02901093
Title: Early Postoperative Imaging of the Labyrinth by Cone Beam CT After Stapes Surgery for Otosclerosis With Correlation to Audiovestibular Outcome
Brief Title: Quantification of Prosthesis Penetration With Conebeam in Otosclerosis
Acronym: QUIPROCOS
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: DAE_2014_15
Record Dates: First submitted 2016-09-07; First posted 2016-09-15 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-03

CONDITIONS: Otosclerosis
Keywords: Stapes surgery; Sensorineural complications; Inner ear; Imaging; Cone Beam CT
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Sensorineural complications of stapes surgery are rare but potentially serious. Imaging is usually performed to identify an underlying cause, such as excessive intravestibular penetration of the prosthesis or pneumolabyrinth suggesting perilymphatic fistula.

Unfortunately, there is very little data in an unselected series of uneventful patients.

The aim of this study is to analyze the depth of prosthesis penetration within the vestibule and the rate of pneumolabyrinth the day or the day after the procedure by performing a Cone Beam CT (CBCT) of the temporal bone in a cohort of unselected patients, and to correlate imaging findings to clinical outcome. This prospective monocentric study is conducted in a tertiary referral medical center. A CBCT is performed in 80 consecutive patients having undergone stapes surgery for otosclerosis, the day or the day after the procedure. Penetration length and location of the prosthesis within the vestibule, as well as presence or absence of a pneumolabyrinth are recorded, and compared to clinical data (vertigo, nystagmus, hearing measurement).

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years old
* patients undergoing stapes surgery for otosclerosis

Exclusion Criteria:

* patient's refusal to participate in the study
* patient under legal protection
* no medical insurance coverage
* pregnant or breast feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing stapes surgery for otosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
location of the medial tip of the prosthesis within the vestibule | 1 day after surgery
  computerized tomography with cone beam
intravestibular length of the prosthesis | 1 day after surgery
  computerized tomography with cone beam
incidence of postoperative pneumolabyrinth | 1 day after surgery
  computerized tomography with cone beam
incidence of vertigo | 1 day after surgery
  clinical assessment
incidence of nystagmus | 1 day after surgery
  clinical assessment
change in pure-tone bone conduction hearing thresholds | between baseline and 1 day after surgery
  measured at 250, 500, 1000, 2000, 3000, 4 000 Hz
Pure-tone audiometry | 7 days, 1 month and 3 months after surgery
bone conduction hearing thresholds | 7 days, 1 month and 3 months after surgery
Speech Discrimination | baseline, 1 month and 3 months after surgery
  audiometry: Speech Discrimination Score at a standard presentation level of 60 decibels (SDS60) expressed in percentages
Speech Reception | baseline, 1 month and 3 months after surgery
  audiometry: Speech Reception Threshold at 50% (SRT50) and/or 100% (SRT100) expressed in dB

REFERENCES:
- [Result] Vandevoorde A, Williams MT, Ukkola-Pons E, Daval M, Ayache D. Early Postoperative Imaging of the Labyrinth by Cone Beam CT After Stapes Surgery for Otosclerosis With Correlation to Audiovestibular Outcome. Otol Neurotol. 2017 Feb;38(2):168-172. doi: 10.1097/MAO.0000000000001306. PMID 28068300